CLINICAL TRIAL: NCT01586065
Title: Use of CGM in Adolescents With Poorly-controlled Type 1 Diabetes
Brief Title: Continuous Glucose Monitoring in Adolescents With Poorly Controlled Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Larry A. Fox, MD, Physician, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R03HD067329-01A1 (NIH)
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; adolescents; poor control; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CGM in adolescents with poorly-controlled T1D (Experimental): Adolescents with poorly controlled type 1 diabetes on insulin pumps were admitted to the clinical research center (CRC) and a continuous glucose sensor was inserted. Sensor glucose (SG) values were compared to plasma glucose measured at least hourly using Yellow Springs Instrument's (YSI) glucose analyzer. SG rather than YSI was used for treatment decisions unless YSI was <70 mg/dL or specific criteria indicating SG and YSI were very discordant were met.
  Interventions: Device: Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — CGM during 24-hr CRC stay.

SUMMARY:
The purpose of this study is to see if children and adolescents with poorly controlled type 1 diabetes will benefit from using a continuous glucose monitor (CGM), a device that can be used to check blood sugars.

DETAILED DESCRIPTION:
Adolescents with type 1 diabetes, HbA1c ≥9% on insulin pumps were admitted to the clinical research center and a continuous glucose sensor was inserted. Sensor glucose (SG) values were compared to plasma glucose measured at least hourly using Yellow Springs Instrument's (YSI) glucose analyzer. SG rather than YSI was used for treatment decisions unless YSI was <70 mg/dL or specific criteria indicating SG and YSI were very discordant were met.

ELIGIBILITY:
Inclusion Criteria:

* 12 to <18 years old
* T1D for at least one year
* Treatment with insulin pump therapy
* A1c ≥9%
* Willingness to comply with study procedures

Exclusion Criteria:

* Current diabetic ketoacidosis
* Hypoglycemia unawareness
* Chronic use of medications that affect recognition of hypoglycemia (e.g., beta blockers)
* Chronic use of medications that mimic symptoms of high or low blood sugars (e.g., decongestants)
* Recent or frequent severe hypoglycemia (2 episodes in the last year; 1 episode in the last 6 months)
* Skin rashes or conditions that may affect CGM placement and wear

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry A Fox, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fox LA, Balkman E, Englert K, Hossain J, Mauras N. Safety of using real-time sensor glucose values for treatment decisions in adolescents with poorly controlled type 1 diabetes mellitus: a pilot study. Pediatr Diabetes. 2017 Jun;18(4):271-276. doi: 10.1111/pedi.12404. Epub 2016 Jul 20. PMID 27435145
- See also: Safety of using real-time sensor glucose values for treatment decisions in adolescents with poorly-controlled type 1 diabetes mellitus: a pilot study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5250611/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Type 1 diabetes, HbA1c ≥9% on insulin pumps
Groups:
- CGM in Adolescents With Poorly Controlled T1D: Adolescents with type 1 diabetes, HbA1c ≥9% on insulin pumps were admitted to the clinical research center and a continuous glucose sensor was inserted. Sensor glucose (SG) values were compared to plasma glucose measured at least hourly using Yellow Springs Instrument's (YSI) glucose analyzer. SG rather than YSI was used for treatment decisions unless YSI was <70 mg/dL or specific criteria indicating SG and YSI were very discordant were met.
Period: Overall Study
Arm/Group | CGM in Adolescents With Poorly Controlled T1D
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adolescents with poorly controlled type 1 diabetes were enrolled.
Groups:
- CGM Use in Adolescents With Poorly Controlled T1D: Adolescents with poorly controlled T1D were admitted to CRC and CGM was placed. The safety of using real-time sensor glucose (SG) data for treatment decisions in adolescents with poorly controlled type 1 diabetes was assessed.
Arm/Group | CGM Use in Adolescents With Poorly Controlled T1D
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 16.3 [15.2 to 17.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of High Glucose Correction Doses Administered.
Description: Principal study outcome was comparing insulin doses using pre- and post-meal sensor versus plasma glucose values. All insulin dose calculations over a 24-hour period were made using sensor glucose concentrations; these doses were compared to the those calculated as if plasma glucose were to be used instead for dose calculations.
Time Frame: 24 hrs
Population: Ten adolescents with poorly controlled type 1 diabetes on insulin pumps were admitted to the clinical research center and a continuous glucose sensor was inserted. Insulin dose calculations based on sensor glucose were compared to calculations made as if based on plasma glucose. 23 paired sensor/plasma glucose values for corrections were analyzed.
Measure: Count of Units; unit: sensor/plasma glucose-based insulin dose
Units Other Than Participants: sensor/plasma glucose-based insulin dose
Groups:
- Insulin Correction Doses Determined Using Sensor Glucose Readings: The insulin doses in this arm were based on calculations using the sensor glucose value.
- Insulin Correction Doses Determined Using YSI Glucose Readings: The insulin doses in this arm were based on calculations using the YSI glucose value.
- All Correction Doses Administered: Insulin correction doses determined using either the sensor or plasma glucose readings
Arm/Group | Insulin Correction Doses Determined Using Sensor Glucose Readings | Insulin Correction Doses Determined Using YSI Glucose Readings | All Correction Doses Administered
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (sensor/plasma glucose-based insulin dose) | 15 | 8 | 23
sensor/plasma glucose-based insulin dose
  Difference between SG and YSI dose calculated (SG-YSI dose) = -2 units | 0 | 2 | 2
  Difference between SG and YSI dose calculated (SG-YSI dose) = -1 unit | 5 | 5 | 10
  Difference between SG and YSI dose calculated (SG-YSI dose) = 0 units | 7 | 1 | 8
  Difference between SG and YSI dose calculated (SG-YSI dose) = +1 unit | 3 | 0 | 3
  Difference between SG and YSI dose calculated (SG-YSI dose) = +2 units | 0 | 0 | 0

2. Secondary Outcome: Pre- and Post-meal (2-3 Hour) Glucose Levels
Description: Mean sensor and plasma pre- and post-meal glucose concentrations for all dinner (n=8), bedtime snack (n=8), and breakfast (n=10) during the study period.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: sensor/plasma glucose levels
Groups:
- Pre- and Post-meal Sensor Glucose Levels: Sensor glucose levels checked before and 2-3 hours after meals
- Pre- and Post-meal Plasma (YSI) Glucose Levels: Plasma glucose levels checked before and 2-3 hours after meals
Arm/Group | Pre- and Post-meal Sensor Glucose Levels | Pre- and Post-meal Plasma (YSI) Glucose Levels
Number analyzed (Participants) | 10 | 10
Number analyzed (sensor/plasma glucose levels) | 26 | 26
mg/dL
  Pre-meal glucose, mean (SD) | 157 (9) | 163 (11)
  Post-meal glucose, mean (SD) | 174 (10) | 183 (12)

ADVERSE EVENTS:
Time Frame: AEs were collected for each participant's admission to the CRC over 24 hrs.
Groups:
- CGM Group: Adolescents using CGM during the CRC admission
Arm/Group | CGM Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGM Group (N=10)
Mild hypoglycemia (Endocrine disorders) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes